CLINICAL TRIAL: NCT04634851
Title: Optimizing Dietary Habits for Kidney Stone Formers Using Telehealth Directed Individualized Nutritional Counseling
Brief Title: Video Home Visits for Dietary Counselling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSFUroVV
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Technology; Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Pilot study comparing intervention (virtual dietary counselling) versus standard of care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): These participants will get virtual home visits with the urologist and dietitian
  Interventions: Behavioral: Virtual home visits
- Control (No Intervention): These participants will get standard urologist and dietitian counseling

INTERVENTIONS:
Behavioral: Virtual home visits — These participants will have a tailored evaluation of dietary choices based on their home dietary environment (refrigerator, pantry, etc). This will be conducted over video exchange.
  Arms: Intervention

SUMMARY:
This pilot study aims to develop a protocol for home video informed dietary counseling with the goal of reducing overall sodium consumption among kidney stone formers. To accomplish this the investigators will: 1)Assess which data available on video visits are most informative to convey patient sodium consumption, and 2) Administer virtual home visits with informed dietary counseling in our intervention arm and compare this to standard dietary counseling looking specifically at the outcome of 24-hour urine sodium excretion results over time. This study will benefit dramatically from the rapid growth of telehealth medical visits as a consequence of the SARS-CoV-2 pandemic, with the ultimate goal to improve and adapt patient dietary counseling for the prevention of kidney stone disease in the new and evolving era of telehealth.

DETAILED DESCRIPTION:
Urolithiasis affects 1 in 11 Americans and is associated with annual health care expenditures of up to $4.5 billion. Fifty percent of stone risk can be attributed to diet and fluid intake. Modifications in sodium intake can dramatically reduce risk of kidney stone disease as determined by 24-hour urine results. Despite this understanding, dietary counseling is largely ineffective as kidney stone formers have difficulty adhering to low sodium diets. The precise reasons behind this are unknown, but it is hypothesized that socioeconomic factors such as low income and low education contribute to a lack of knowledge of, and access to, healthy alternatives to salty foods. The relationship between lithogenic diet consumption and stone disease requires a more in depth understanding of patients' home food environments, dietary habits, and perceived barriers to following a low-sodium diet. This understanding will help direct appropriate interventions to prevent recurrent stones.

Routine historic face-to-face clinic visits rapidly have been replaced with telehealth encounters with the SARS-CoV-2 pandemic. Such changes will likely remain the standard of care and will define the new "normal" for some time. This presents an opportunity to integrate robust information now available through the exponential growth of video visits with directed dietary counseling. Through video exchange with patients in their homes an abundance of previously untapped information is immediately available to healthcare providers. Smartphone video capabilities are available to most stone patients irrespective of their financial status. Images from telehealth video visits, including patient lifestyle, behaviors, resources, and home environment will give objective data as to types of food consumed regularly by patients and their capacity to prepare healthy foods at home.

The following specific aims are proposed: 1) Assess which data from video visits are most informative for identifying how to counsel patients to reduce patient sodium intake, and 2) Administer virtual home visit-informed individualized dietary counseling to stone formers and compare this to survey-informed dietary counseling. 24-hour urinary sodium results and patient dietary sodium knowledge and perceptions will be monitored over 6 months. This study will leverage the rapid growth of telehealth medical visits as a consequence of the SARS-CoV-2 pandemic to better understand and improve food consumption behavior of recurrent stone formers.

ELIGIBILITY:
Inclusion Criteria:

* Patients known to have a history of calcium-based kidney stone disease verified by stone analysis (stones containing calcium oxalate(CaOx) or calcium phosphate(CaP) on stone analysis), or patients with a diagnosis of kidney stone disease verified by imaging (computerized tomography, ultrasound, or plain film/x-ray) and a prior 24-hour urine results with elevated SS CaOx>8 or SS CaP>1.25.
* Patients 18 years or older.
* Patients with a smartphone, internet capable tablet, or video capable laptop.
* Patients with a household member with a smartphone, internet capable tablet, or video capable laptop.

Exclusion Criteria:

* Pregnant patients.
* Patients unable to produce a urine sample.
* Patients who have previous surgical reconstruction involving incorporation of bowel in the urinary tract.
* Patients with known sodium regulation abnormalities (adrenal tumors, pituitary tumors, glucocorticoid deficiency, hypothyroidism, syndrome of inappropriate antidiuretic hormone secretion, nephrotic syndrome, severe congestive heart failure, severe hepatic impairment, etc.).
* Patients on medications significantly affecting urinary sodium levels (lithium, amphotericin, vasopressin V2-receptor antagonists, lactulose, for example).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinary sodium | baseline, 12 weeks, 24 weeks
  24hr urinary sodium, mean change in mmol/24hrs of excreted urinary sodium from baseline over 24 weeks (Three time points will be recorded: baseline, after 12 weeks, after 24 weeks. Outcome will be mean change from baseline. We will take the average of change from baseline at 12 weeks and change from baseline at 24 weeks)

SECONDARY OUTCOMES:
Food Frequency Questionnaire (FFQ) | baseline, 12 weeks, 24 weeks
  Change in response to NutritionQuest® block sodium screener Food Frequency Questionnaire (FFQ), (Three points will be recorded: baseline, after 12 weeks, after 24 weeks. Outcome will be change from baseline over time. We will look specifically for a reduction in self reported weekly consumption of high sodium foods including soups, pizza, hot dogs, lunch meets, table salt, cooking salt, etc. Results will be noted for change from baseline at 12 weeks and at 24 weeks)
Short Sodium Knowledge Survey (SKSS) | baseline, 12 weeks, 24 weeks
  Change in response to Short Sodium Knowledge Survey (SKSS), (Three points will be recorded: baseline, after 12 weeks, after 24 weeks. Outcome will be change from baseline over time. We will look specifically for a an increased frequency in accurate identification of high sodium foods and accurate identification of dietary sodium intake recommendations. Results will be noted for change from baseline at 12 weeks and at 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: David Bayne, MD, MPH, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD